CLINICAL TRIAL: NCT04487431
Title: Single-center, Open-label, Non-placebo-controlled, Single-dose Study in Healthy Male Participants to Determine the Pharmacokinetics of BAY 1817080 Oral Solution (Part A) and to Investigate the Pharmacokinetics, Metabolic Disposition and Mass Balance of [14C]BAY 1817080 Oral Solution (Part B)
Brief Title: A Trial to Learn How a New Liquid Form of BAY1817080 is Tolerated and Taken up by the Body of Healthy Male Participants (Part A). By Labeling BAY1817080 With a Radioactive Substance (Carbon 14) Researchers Want to Learn How the Study Drug is Processed and Excreted by the Body After Dosing (Part B)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20330; 2020-000519-54 (EudraCT Number)
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Endometriosis Related Pain; Overactive Bladder; Diabetic Neuropathic Pain; Refractory or Unexplained Chronic Cough
Keywords: Healthy volunteers; Pharmacokinetics (PK)
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY1817080 Part A (Experimental): Healthy male participants will receive BAY1817080 given as an oral solution (study Part A)
  Interventions: Drug: BAY1817080
- [14C]BAY1817080 Part B (Experimental): Healthy male participants will receive BAY1817080 blended with [14C]BAY1817080 given as an oral solution (study Part B).
  Interventions: Drug: [14C]BAY1817080

INTERVENTIONS:
Drug: BAY1817080 — Oral single dose
  Arms: BAY1817080 Part A
Drug: [14C]BAY1817080 — Oral single dose
  Arms: [14C]BAY1817080 Part B

SUMMARY:
Researchers are looking for a new way to treat people suffering either from a condition where the bladder is unable to hold urine normally (overactive bladder), or a condition in which tissue similar to the tissue that normally lines the inside of the womb grows outside the womb (endometriosis) or a condition where the cough lasts longer than 8 weeks in adults (chronic cough). BAY1817080 is a new drug that is in development as a potential treatment for these conditions.

In this trial, the researchers want to learn how a new liquid form of BAY1817080 is taken up by the body in a small number of healthy participants. The trial will include men who are aged 18 to 54.

The trial will have 2 parts: A and B. The participants in Part A will stay at the trial site for about 5 days. During this time, the participants will take 1 dose of a liquid form of BAY1817080 by mouth. The doctors will take blood and urine samples and check the participants' health. Part A will be done so the researchers can see how much BAY1817080 gets into the participants' blood. The participants in Part B will stay at the trial site for about 16 days followed by a maximum of 4 re-admission visits over 24 hours at intervals of 7 days. These participants will take 1 dose of a liquid form of BAY1817080 labeled with a radioactive substance (carbon 14), which means it is "radiolabeled". This allows the researchers to understand how BAY1817080 moves through and leaves the body. During Part B, the doctors will take blood, urine, stool, and vomit samples if applicable. They will also check the participants' health.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent as described in Appendix which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol;
* Ability to understand and follow study-related instructions;
* Participant has signed the ICF before any study specific tests or procedures are done;
* Healthy male participant;
* Age: 18 to 54 years (inclusive) at the time of informed consent and first dose of study medication;
* Body mass index (BMI) ≥18 and ≤30 kg/m^2 at Screening;
* Body weight of at least 45 kg at Screening;
* Participant agrees to use contraception as described in Appendix.

Exclusion Criteria:

* Presence or history of clinically relevant cardiovascular, central nervous system (CNS), hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash;
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations);
* Known severe allergies, e.g., allergies to more than 3 allergens, allergies affecting the lower respiratory tract (e.g., allergic asthma), allergies requiring therapy with corticosteroids or significant nonallergic drug reactions;
* Febrile illness within 1 week before study drug administration;
* Current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent occurrence of heartburn [more than once per week], or any gastrointestinal surgical intervention [e.g. cholecystectomy]);
* Participant has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Screening;
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of study intervention will not be normal;
* Poor peripheral venous access;
* Regular use of medicines within 14 days prior to administration of study intervention;
* Regular use of therapeutic or recreational drugs, e.g., cannabis, carnitine products, anabolics, high dose vitamins within 3 months prior to screening;
* Any use of medicines or substances within 14 days prior to administration, which oppose the study objectives or might affect the PK of BAY1817080 (e.g., laxatives, loperamide, metoclopramide, antacids, H2-receptor antagonists, systemic antibiotics, CYP3A4 inducers, CYP3A4 inhibitors, "organic anion transporting polypeptide" (OATP) / "breast cancer resistance protein" (BCRP) substrates, P-gp substrates and inhibitors). Relevant medication of individual participants will be discussed with the study medical expert before first dosing in the study.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
AUC of BAY1817080 in plasma (Part A) | Pre-dose, post-dose on Day 1 (up to 16 hours), Days 2 to 4 (every 12 hours)
  Area under the concentration vs. time curve
Maximum observed concentration of BAY1817080 in plasma (Cmax) (Part A) | Pre-dose, post-dose on Day 1 (up to 16 hours), Days 2 to 4 (every 12 hours)
Radioactivity excreted in urine of BAY1817080 and its metabolites as a percentage of the dose (%AE,ur) (Part B) | Pre-dose, Day 1 (0-12 h and 12-24 h), Days 2 to 15, 22, 29, 36, 43
Radioactivity excreted in feces of BAY1817080 and its metabolites as a percentage of the dose (%AE,fec) (Part B) | Pre-dose, Days 1 to 15, 22, 29, 36, 43
Radioactivity excreted in vomit (if applicable) of BAY1817080 and its metabolites as a percentage of the dose (%AE,v) (Part B) | Up to 12 hours post-dose
Whole blood to plasma ratio of total radioactivity (Part B) | Pre-dose, post-dose on Day 1 (up to 12 hours), Days 2 to 10, 12, 15, 22, 29, 36, 43
AUC of [14C]BAY1817080 in Plasma (Part B) | Pre-dose, post-dose on Day 1 (up to 12 hours), Days 2 to 10, 12, 15
Cmax of [14C]BAY1817080 in plasma (Part B) | Pre-dose, post-dose on Day 1 (up to 12 hours), Days 2 to 10, 12, 15
AUC of total radioactivity (Part B) | Pre-dose, post-dose on Day 1 (up to 12 hours), Days 2 to 10, 12, 15, 22, 29, 36, 43
Cmax of total radioactivity (Part B) | Pre-dose, post-dose on Day 1 (up to 12 hours), Days 2 to 10, 12, 15, 22, 29, 36, 43

SECONDARY OUTCOMES:
Number of participants with Treatment-emergent adverse events (TEAEs) (Part A) | From first dose up to Day 15
Number of participants with maximum severity of TEAEs (Part A) | From first dose up to Day 15
Number of participants with TEAEs (Part B) | From first dose up to Day 15
Number of participants with maximum severity of TEAEs (Part B) | From first dose up to Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- PRAHealthSciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Reif S, Schultze-Mosgau MH, Engelen A, Piel I, Denner K, Roffel A, Tiessen R, Klein S, Francke K, Rottmann A. Mass Balance and Metabolic Pathways of Eliapixant, a P2X3 Receptor Antagonist, in Healthy Male Volunteers. Eur J Drug Metab Pharmacokinet. 2024 Jan;49(1):71-85. doi: 10.1007/s13318-023-00866-0. Epub 2023 Dec 3. PMID 38044419